CLINICAL TRIAL: NCT00888173
Title: A Phase II Evaluation of Brivanib (BMS582664), an Oral, Multitargeted Growth Factor Tyrosine Kinase Inhibitor in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Brivanib Alaninate in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0229I; NCI-2011-01918 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CA182-029; CDR0000641191; GOG-0229I (Other: NRG Oncology); GOG-0229I (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-08

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Adenocarcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Endometrial Transitional Cell Carcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brivanib alaninate) (Experimental): Patients receive brivanib alaninate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brivanib Alaninate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Brivanib Alaninate — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well brivanib alaninate works in treating patients with endometrial cancer that has come back (recurred) or is persistent. Brivanib alaninate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of brivanib (brivanib alaninate) for patients with recurrent or persistent endometrial cancer with the frequency of patients who survive progression-free for at least 6 months after initiating therapy or have objective tumor response..

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival. II. To determine the nature and degree of toxicity of brivanib as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v)3.0 in this cohort of patients.

TERTIARY OBJECTIVES:

I. To determine whether activating mutations in fibroblast growth factor receptor 2 (FGFR2) are associated with progression-free survival status > 6 months following brivanib treatment, objective tumor response following brivanib treatment, or endometrioid histology.

II. To explore the associations between select biomarkers and response to brivanib (progression-free survival status > 6 months and objective tumor response), measures of clinical outcome (progression-free survival and overall survival) or disease status including histologic cell type: i) mutations in FGFR2 or phosphatase and tensin homolog (PTEN) in deoxyribonucleic acid (DNA) from formalin-fixed and paraffin-embedded (FFPE) tumor or normal blood cells; ii) immunohistochemical (IHC) expression of the FGFR family and ligands, steroid receptor isoforms or phosphorylated (p) v-akt murine thymoma viral oncogene homolog 1 (AKT) in FFPE tumor; iii) concentration or the change in the concentration of vascular endothelial growth factor (VEGF) or type IV collagen in pre-cycle 1, pre-cycle 2 and/or pre-cycle 3 plasma.

III. To explore the relationship among the panel of biomarkers evaluated in this cohort: i) mutations in FGFR2 or PTEN; ii) IHC expression of the FGFR family and ligands, steroid receptor isoforms or pAKT; iii) concentration or the change in the concentration of VEGF or type IV collagen.

OUTLINE:

Patients receive brivanib alaninate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required

  * Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell, and transitional cell carcinoma
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Patients must have at least one ?target lesion? to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST); tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III or Rare Tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer will be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent endometrial disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
  * Note: Patients on this non-cytotoxic study are allowed to receive one additional cytotoxic chemotherapy regimen for management of recurrent or persistent endometrial disease, as defined above; however, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
* Patients must NOT have received any non-cytotoxic therapy for management of endometrial cancer with the exception of hormonal therapy
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to Common Terminology Criteria (CTCAE v3.0) grade 1
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin > 9 g/dl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v3.0 grade 1
* Urinalysis needs to be assessed at baseline and proteinuria must be less than or equal to 3+ by dipstick (CTCAE v3.0 grade 2 or less); if the urine dipstick is > 3+, a 24-hour protein level can be done, as clinically indicated by the investigator; the 24-hour protein level must be less than or equal to 3.5 g/24 hours (CTCAE v3.0 grade 2 or less)
* Bilirubin less than or equal to 1.5 x ULN (CTCAE v3.0 grade 1)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Albumin greater than or equal to 2.5 g/dl
* Neuropathy (sensory and motor) less than or equal to CTCAE v3.0 grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is < 1.5 x ULN; patients on therapeutic warfarin are excluded from trial, anticoagulation with low molecular weight heparin is allowed
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test performed 48 hours prior to study entry and be practicing an effective form of contraception during the study and for at least 3 months after receiving the final treatment of brivanib
* All patients must have a baseline electrocardiogram completed prior to study entry; baseline electrocardiogram (ECG) should be repeated if corrected QT interval (QTc) is found to be > 450 msec; QTc must NOT be > 450 msec on both ECGs performed during the same visit

Exclusion Criteria:

* Patients who have had prior therapy with brivanib or anti-vascular, anti-PDGFR (platelet-derived growth factor receptor) or anti-FGFR (fibroblast growth factor receptor) therapy
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted below, are excluded if there is any evidence of the other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients that are on required chronic anti-platelet therapy (aspirin > 300 mg/day, or clopidogrel greater than or equal to 75 mg/day)
* Patients with gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE grade >= 3 within 30 days prior to study entry
* Patients with a history of poor wound healing, non healing ulcers or bone fractures within the last 3 months
* Patients with uncontrolled or significant cardiovascular disease including:

  * Myocardial infarction within 12 months
  * Uncontrolled angina within 12 months
  * Class III-IV New York Heart Association (NYHA) congestive heart failure
  * Uncontrolled hypertension (systolic blood pressure [BP] > 150 or diastolic BP > 100 mmHg for 24 hours) despite optimized anti-hypertensive therapy; BP must be below 150/100 mmHg at screening; subjects with a history of hypertension who are receiving treatment with calcium channel blockers that are cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors should be changed to an alternative antihypertensive medication before study entry
  * History of stroke, transient ischemic attack (TIA), or other central nervous system (CNS) ischemic event
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Patients must have pre-therapy left ventricle ejection fraction (LVEF) testing and have an ejection fraction > 50%
  * Patients with valvular heart disease >= CTCAE grade2
* Patients with a serious uncontrolled medical disorder or active infection which would impair the ability of the subject to receive protocol therapy or whose control may be jeopardized by the complications of this therapy
* Pre-existing thyroid abnormality with thyroid function that can not be maintained in the normal range with medication
* Patients with hyponatremia (sodium < 130 mEq/L)
* Patients with active/known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Patients with known brain metastases
* Patients who are pregnant or nursing
* Patients with inability to swallow tablets or untreated malabsorption syndrome
* Baseline serum potassium < 3.5 mmol/L (potassium supplementation may be given to restore the serum potassium above this level prior to entry study)
* Patients on therapeutic warfarin anticoagulation will be excluded; patients converted to anticoagulation with a heparin compound will be allowed provided the patient?s PT is such that international normalized ratio (INR) is =< 1.5 x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-07-06 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Powell, Principal Investigator — NRG Oncology
Locations (35):
- United States (35):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 7/6/2009 and suspended to accrual on 12/14/2009. The study reopened on 9/7/2010 and closed on 1/3/2011.
Groups:
- Brivanib: Brivanib 800 mg orally every day (one cycle = 28 days) until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Brivanib
Started | 45
Completed | 43
Not Completed | 2
Not completed — Wrong Primary | 1
Not completed — Ineligible: required test not done | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brivanib
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 3
  50-59 years | 12
  60-69 years | 15
  70-79 years | 11
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival > 6 Months
Description: Whether or not the patient survived progression-free for at least 6 months.
Time Frame: For patients whose disease can be evaluated by physical examination, progression was assessed prior to each cycle for 6 months.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Brivanib
Number analyzed (Participants) | 43
percentage of participants | 30.2 [19 to 44]

2. Primary Outcome: Tumor Response
Description: Per response evaluation criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30 % decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: If evaluated by physical exam, response was assessed prior to each cycle. If evaluated by CT or MRI, response was assessed during course of therapy. Overall time frame is up to 6 months.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Brivanib
Number analyzed (Participants) | 43
percentage of participants | 18.6 [9 to 31]

3. Secondary Outcome: Duration of Overall Survival
Description: Characterized graphically with Kaplan-Meier estimates and using descriptive statistics. The effect of cell type (type I versus type II endometrial cancers) on overall survival will be examined.
Time Frame: From entry into the study to death or the date of last contact, assessed up to 5 years
Population: Eligible and Treated Patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Brivanib
Number analyzed (Participants) | 43
months | 10.7 [9.2 to 18.1]

4. Secondary Outcome: Duration of Progression-free Survival
Description: Characterized graphically with Kaplan-Meier estimates and using descriptive statistics. The effect of cell type (type I versus type II endometrial cancers) on progression-free survival will be examined.
Time Frame: Form study entry until disease progression, death or date of last contact, assessed up to 5 years
Population: Eligible and Treated Patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Brivanib
Number analyzed (Participants) | 43
months | 3.3 [2.0 to 3.8]

5. Secondary Outcome: Severity of Adverse Events as Assessed by CTCAE v3.0 Criteria
Description: Adverse Events (grade 3 or higher)
Time Frame: Up to 5 years
Population: Eligible and Treated Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Brivanib
Number analyzed (Participants) | 43
Participants
  Leukopenia | 1
  Anemia | 2
  Cardiac | 9
  Coagulation | 5
  Constitutional | 2
  Dermatologic | 1
  Gastrointestinal | 12
  Genitourinary/Renal | 1
  Infection | 2
  Lymphatics | 2
  Metabolic | 10
  Musculoskeletal | 2
  Other Neurological | 4
  Pain | 4
  Vascular | 2
  Death, Not CTC coded | 2

6. Other Pre Specified Outcome: Activating Mutation in FGFR2
Description: Will be correlated with clinical measures of outcome such as tumor response, progression-free survival (PFS), and endometrioid histology.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Concentration of VEGF and Type IV Collagen
Description: Will be correlated with PFS, OS, tumor response, and histologic cell type.
Time Frame: Baseline to up to pre-course 3
Reporting Status: Not Posted

8. Other Pre Specified Outcome: IHC Expression of FGFR Family and Ligands, Steroid Receptor Isoforms, and pAKT
Description: Will be correlated with PFS, OS, tumor response, and histologic cell type.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mutations in FGFR2 and PTEN
Description: Will be correlated with PFS, overall survival (OS), tumor response, and histologic cell type.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment
Arm/Group | Brivanib
Serious Adverse Events (participants affected / at risk) | 18/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brivanib (N=43)
Hypertension (Cardiac disorders) | 2
Inr (Vascular disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Mental Status (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Pain: Tumor (General disorders) | 1
Obstruction, Gu - Bladder (Renal and urinary disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brivanib (N=43)
Rhinitis (Immune system disorders) | 3
Otitis Middle Ear (Ear and labyrinth disorders) | 1
Otitis External Ear (Ear and labyrinth disorders) | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 4
Platelets (Blood and lymphatic system disorders) | 10
Leukocytes (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 21
Palpitations (Cardiac disorders) | 2
Ventricular Arrhythmia - Fibrillation (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 13
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 2
Cardiac General - Other (Cardiac disorders) | 1
Inr (Vascular disorders) | 5
Ptt (Vascular disorders) | 2
Constitutional Symptoms - Other (General disorders) | 1
Fever (General disorders) | 1
Weight Loss (General disorders) | 6
Fatigue (General disorders) | 28
Insomnia (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 4
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 5
Induration (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 2
Hand-Foot (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 3
Dental: Teeth (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 5
Distention (Gastrointestinal disorders) | 2
Incontinence, Anal (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 9
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 11
Anorexia (Gastrointestinal disorders) | 19
Dehydration (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 27
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 19
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 4
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bone (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Infection - Other (Infections and infestations) | 2
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 3
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 3
Inf W/Gr 3 Or 4 Anc: Bone (Osteomyelitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: External Ear (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 4
Ast (Metabolism and nutrition disorders) | 22
Gfr (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Alt (Metabolism and nutrition disorders) | 22
Alkaline Phosphatase (Metabolism and nutrition disorders) | 14
Bilirubin (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 13
Hyperuricemia (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 2
Fracture (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Psychosis (Nervous system disorders) | 2
Mood Alteration - Euphoria (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 3
Mood Alteration - Anxiety (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Speech Impairment (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 3
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 9
Neuropathy,cranial - Cn Xii Motor-Tongue (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 14
Neuropathy-Motor (Nervous system disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Pain: Pelvis (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Chest Wall (General disorders) | 2
Pain: Throat/Pharynx/Larynx (General disorders) | 2
Pain: Head/Headache (General disorders) | 15
Pain: Extremity-Limb (General disorders) | 7
Pain: Back (General disorders) | 9
Pain: Joint (General disorders) | 6
Pain: Kidney (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Oral Cavity (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 11
Pain: Skin (General disorders) | 1
Pain: Middle Ear (General disorders) | 2
Pain: External Ear (General disorders) | 2
Pain: Liver (General disorders) | 1
Pain: Muscle (General disorders) | 2
Pain: Neuralgia (General disorders) | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Perforation, Gu - Bladder (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 3
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No